## **Informed Consent Form**

Trial Title: An open-label, multi-center first in human, dose escalation, and

cohort expansion phase I clinical trial to evaluate the safety,

tolerability, pharmacokinetic characteristics and and efficacy of

DXC006 in patients with advanced solid tumors and hematologic

malignancies.

Sponsor: Hangzhou DAC Biotechnology Co., Ltd.

Version number: 1.2

Version Date: October 30, 2023

Name of patient

Participant Number:

Note: when applying this template, corresponding modifications should be made according to the different study contents.

# Informed Consent Form · Informed Consent Page Dear patient:

The doctor has diagnosed you with solid tumors and hematomas, including but not limited to small cell carcinoma of lung, multiple myeloma, neuroblastoma. We will invite you to participate in an open-label, multi-center, first-in-human Phase I clinical study to evaluate the safety, tolerability, pharmacokinetic profile and efficacy of DXC006 in the clinical treatment of patients with multiple solid tumors, including small cell carcinoma of lung, multiple myeloma, and neuroblastoma. This study is a domestic multicenter Phase I clinical project, Study No.: DXC006-001. This protocol has been reviewed and agreed by the Ethics Committee of Cancer Center of Sun Yat-sen University.

Please read the following as carefully as possible before you decide whether to take part in this study. It can help you understand the study and why it is being conducted, the procedures and duration of the study, and the possible benefits, risks, and discomforts that may result from taking part in the study. If you wish, you can also discuss it with your relatives and friends, or ask your doctor for an explanation to help you make a decision.

#### I. Study Background and Study Objectives

#### 1.1 Disease Burden and Treatment Status

Usually, a four-part structure can be used: (1) an overview of health problems or research questions: definition of health problems, epidemiological data, etiology, natural history of diseases, disease burden, etc.; (2) Scientific hypothesis: mechanism or principle; (3) Clinical application, e.g., treatment research needs to explain the treatment method; (4) There is currently available evidence on the necessity of the study to explain why this study should be conducted.

Malignant neoplasms are a major public health problem worldwide, while China has the highest number of new cases and deaths in the world, far exceeding the rest of the world. Lung cancer is the most common malignant tumor with the fastest increase in incidence in China in the past 30 years. It is estimated that 2.2 million new cases and 1.79 million deaths each year are the leading cause of cancer-related deaths worldwide, with Small Cell Carcinoma of Lung (SCLC) accounting for approximately 15% of lung cancer cases. Multiple myeloma (MM), the second most common malignancy of the hematological system, is a malignant disease with abnormal proliferation of clonal plasma cells,

accounting for 10% of all hematological malignancies and 1-1.8% of all cancers. Neuroblastoma (NB), the most common extracranial solid tumor in childhood, is derived from undifferentiated sympathetic ganglion cells. Therefore, tumors can occur in any location with embryonic sympathetic ganglion cells, accounting for  $8\% \sim 10\%$  of childhood malignant tumors, with a mortality rate of 15%. Its diversity biological behavior, complex etiology, and tumor heterogeneity is more obvious, which brings a great challenge for clinical treatment.

Antibody Drug Conjugate (ADC) has scientifically utilized the specificity and high affinity of monoclonal antibodies to cancer cell surface targets and the powerful lethality of small molecule cytotoxic compounds, and the specific function of linkers in the targeted release of chemotherapeutic drugs in cancer cells has been one of the hottest in the field of tumor precision therapy in recent years.

The drug DXC006 independently developed by Hangzhou DAC Biotechnology Co., Ltd. The proposed indications for DXC006 are small cell carcinoma of lung, multiple myeloma, neuroblastoma and other solid tumors and hematomas. DXC006 showed significant anti-tumor activity and good safety in preclinical animal studies.

DXC006 is the investigational product used in this study. The investigational drug has been approved by the National Medical Products Administration (NMPA) to conduct clinical trials in China, but has not been approved for marketing. We are investigating whether DXC006 is effective in a variety of solid tumors such as small cell carcinoma of lung, multiple myeloma, neuroblastoma, and hematomas.

#### 1.2 Objectives

**Primary Study Objectives** 

• To evaluate the safety and tolerability of DXC006 in patients with various solid tumors and hematomas such as small cell carcinoma of lung, multiple myeloma and neuroblastoma, determine the Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT) of DXC006, and determine the Recommended Dose (RP2D) for phase II clinical trials.

Secondary Study Objectives

- To evaluate the pharmacokinetic (PK) characteristics of DXC006 in patients with various solid tumors, such as small cell carcinoma of lung, multiple myeloma and neuroblastoma;
- To evaluate the immunogenicity of DXC006 in patients with various solid tumors and hematomas such as small cell carcinoma of lung, multiple myeloma and neuroblastoma;
- To preliminarily evaluate the clinical efficacy of DXC006 in patients with various solid

tumors and hematomas such as small cell carcinoma of lung, multiple myeloma and neuroblastoma;

**Exploratory Objectives** 

- To explore the major metabolites of the drug in humans.
- To investigate the correlation between the expression level of biomarkers in tumor tissue and the therapeutic effect.

#### 1.3 Number of Study Participants and Expected Participants

This study is a multi-center, open-label, dose-escalation and expanded enrollment phase I clinical study. The leading unit is the Cancer Center of Sun Yat-sen University, and the participating center is Hunan Cancer Hospital. The exploratory study is divided into two phases: dose escalation and dose expansion. Up to approximately 50 patients with small cell carcinoma of lung and multiple myeloma are planned to be enrolled in the dose escalation phase. The dose expansion enrollment phase is to select an appropriate dose for the study based on the previous safety and preliminary efficacy assessments, and approximately 20-60 patients are planned to be enrolled.

#### II. Unsuitable participants

#### **Exclusion Criteria**

Note the relationship between inclusion and exclusion criteria: inclusion criteria define the subject of the study and determine the representation of the study population; exclusion criteria define the individuals in the subject of the study that may affect the study and determine the homogeneity of the study population.

Patients will not be included in the study if they meet any of the following criteria:

- 1. Received plasma exchange; use > 10 mg daily of prednisone for more than 3 consecutive days or equivalent systemic corticosteroid therapy or equivalent anti-inflammatory active medication within 14 days prior to the first dose (for short-term use to prevent contrast allergy, enrollment may be included);
- 2. Received systemic anti-myeloma therapy or study drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose; Received radiotherapy within 14 days prior to the first dose;
- 3. Received monoclonal antibody treatment within 30 days prior to the first dose;
- 4. Received autologous hematopoietic stem cell transplantation within 100 days prior to the first dose;

- 5. Received allogeneic hematopoietic stem cell transplantation (HSCT) or with a history of solid organ transplantation;
- 6. Received related therapy (limited to Phase Ia clinical trials);
- 7. With symptomatic brain or meningeal metastases; stable central nervous system involvement may be enrolled (no evidence of radiographic progression, central nervous system symptoms, and no need for steroids and anticonvulsant therapy for at least 1 month prior to the first dose) and any neurological symptoms have returned to baseline. All patients at screening should have brain CT/MRI performed prior to study entry.
- 8. With symptomatic amyloidosis, active plasma cell leukemia, active POEMS syndrome at screening;
- 9. With evidence of cardiovascular risk, including any of the following:
- a.QTcF interval  $\geq$  470 milliseconds (QT interval should be corrected for heart rate using Fridericia's formula [QTcF]);
- b. With evidence of currently clinically significant untreated arrhythmias, including clinically significant electrocardiographic abnormalities such as 2nd-degree (Mobitz type II) or 3rd-degree atrioventricular (AV) block.
- c. With history of myocardial infarction, acute coronary syndrome (including unstable angina), coronary angioplasty or stenting or bypass grafting within 6 months prior to screening.
- d. With class III or IV heart failure defined by the New York Heart Association functional classification system;
- e. With uncontrolled severe hypertension (systolic blood pressure  $\geq$  160 mmHg or diastolic blood pressure  $\geq$  100 mmHg);
- 10. With dyspnoea or current need for continuous oxygen therapy, or current active pneumonia or interstitial lung disease (except mild as judged by the investigator);
- 11. With history of other primary malignancies, with the following exceptions: malignancies that have been cured and have a very low risk of recurrence within 5 years, such as basal cell carcinoma of the skin and squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast;
- 12. With severe unhealed wound ulceration or fracture, or major surgery within 28 days prior to administration or expected major surgery during the clinical study;
- 13. Allergy to any component or excipient of DXC006 (sodium citrate, citric acid, sucrose, polysorbate 20 (for injection));

- 14. With active hepatitis B (HBV-DNA greater than the upper limit of central normal or HBV-DNA greater than 1000 copies/mL); hepatitis C infection (positive for hepatitis C antigen or positive result of hepatitis C RNA PCR).
- 15. With Known human immunodeficiency virus (HIV) seropositivity; active syphilis (only syphilis antibody positive can be enrolled); possible active tuberculosis (chest imaging within 3 months prior to the first dose suggests active tuberculosis infection); 16. With active bleeding within 30 days prior to screening, or at risk of major
- 16. With active bleeding within 30 days prior to screening, or at risk of major gastrointestinal bleeding and hemoptysis as judged by the investigator; or hereditary bleeding tendency or coagulation dysfunction, or bleeding symptoms requiring other medical intervention;
- 17. With serious arterial/venous thrombotic events, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism, within 6 months prior to study drug administration;
- 18. Female subjects with a positive serum pregnancy test or breastfeeding;
- 19. With active infection requiring medical treatment (CTCAE Grade  $\geq$  2); uncontrollable pleural effusion, ascites, pericardial effusion requiring repeated drainage;
- 20. Received live attenuated vaccine within 28 days prior to the first dose;
- 21. With other conditions that, as judged by the investigator and the sponsor, may affect the patient's participation in this study.

#### III. What will be required if participating in the study?

- 1. Before you are enrolled in the study, your doctor will ask and record your medical history and assess the patient's condition. If the inclusion criteria are met and you voluntarily participate in the study, you will sign the informed consent form. If you do not want to participate in the study, it will not lead to prejudice against you or affect your medical care.
- 2. If you volunteer to participate in the study, the following steps will be followed:

You will complete further detailed tests under the guidance of the study doctor after you sign the informed consent form. The study doctor will judge whether you meet the inclusion and exclusion criteria in the protocol based on the results of your tests to decide whether you can continue in the study.

Screening Visit

The study doctor will ask about your demographic information as well as specific information about your medical history, including your prior treatment history (including

chemotherapy, biotherapy, immunotherapy and targeted therapy, or all relevant anti-tumor therapies) and how cancer responds to these treatments and drugs;

- · Laboratory tests: serum virological testing with approximately 3-5 mL of blood collection required;
- · Evaluate heart function with color echocardiography or multi-gated acquisition (MUGA) scans;
- · The study doctor will make an initial assessment of your disease by evaluating the results of your previous tests to confirm whether you have a bone marrow aspirate;
- · The study doctor will evaluate your previous results to confirm whether target immunohistochemistry and relevant genetic testing will be performed on you;
- The study doctor will assess your previous results to confirm whether you have imaging studies (whole-body X-ray, local or whole-body CT, local or whole-body MRI, or PET-CT);
- · If you have a history of extramedullary plasmacytoma or have relevant clinical symptoms, the study doctor will evaluate your previous test results to confirm if a plasmacytoma test (CT or MRI) is performed.

To be completed within 7 days prior to the first dose:

- · Physical examination: including physical examination, height, weight, vital signs (heart rate/blood pressure/respiration/body temperature), performance status, etc.;
- Laboratory tests: including blood tests: hematology, blood biochemistry, coagulation function, and one or more of the following if necessary: serum immunoglobulin quantification, serum protein electrophoresis, serum free light chain, serum immunofixation electrophoresis, β2 microglobulin, corrected serum calcium, urine VMA, serum NSE, pregnancy test for women of childbearing potential, and the blood volume required for blood test is about 10-20 mL; Urinalysis: urine routine, and 24-hour urine protein electrophoresis and urine immunofixation electrophoresis if necessary, with a urine sample collection volume of approximately 10 mL; Fecal routine: including fecal occult blood, stool samples collected about the size of soybeans.
  - · An electrocardiogram to assess the electrical activity of your heart;

#### Treatment Visit

If you have completed all the tests at screening and have been confirmed by the study doctor that you are suitable for this study, you will enter the appropriate dose group in the order in which the screening examinations are completed, and the study drug will be administered by intravenous infusion, and the corresponding tests will be performed at the same time. If laboratory parameters or other test results are abnormal during the study, the investigator may increase the number of tests or perform further tests as clinically indicated and record them at

unscheduled visits. You will complete the appropriate tests at different time points during the treatment period, including but not limited to the following:

#### ① Cycle 1

You will need to be admitted to the study ward the day before starting the medication and continue until after the 2nd dose or as deemed appropriate by the study doctor. The study doctor will ask you questions about any symptoms, diseases, and drug changes that you have experienced since the Screening Visit.

Cycle 1 Day 1:

You will receive an intravenous infusion of DXC006 on Cycle 1 Day 1.

Before administration, you need to cooperate to complete the following items:

Vital signs, weight, physical examination, performance status assessment, electrocardiogram, and 7 ml of blood sample for study drug concentration monitoring; Collect approximately 3.5 ml of blood sample for immunogenicity testing;

Laboratory tests: including blood tests (hematology, coagulation function, etc.), and the blood sampling volume required for blood test is about 10-20 mL; Urinalysis, urine sample collection volume of approximately 10 mL; Fecal routine, stool samples are collected approximately the size of soybeans. If these tests are obtained within 3 days prior to the first dose at screening, they do not need to be repeated.

After administration, you need to cooperate to complete the following items:

Vital signs are monitored, electrocardiograms are performed, and approximately 7 mL of blood samples are collected for study drug concentration monitoring;

Cycle 1 Day 2

Vital signs, physical examination, electrocardiogram, and approximately 7 mL of blood will be collected for study drug concentration monitoring.

Cycle 1 Day 3

Vital signs are monitored, physical examination, and ECG are performed.

Cycle 1 Day 4

Approximately 7 mL of blood samples are collected for study drug concentration monitoring.

Cycle 1 Day 8:

Vital signs are monitored, physical examination, and ECG are performed.

Laboratory tests: including blood tests (hematology, blood biochemistry, coagulation function), and the required blood collection volume is about 10-20 mL; Urine routine, urine sample collection volume is approximately 10 mL. Approximately 7 mL of blood samples will

also be collected for study drug concentration monitoring.

Cycle 1 Day 11:

Approximately 7 mL of blood samples are collected for study drug concentration monitoring.

Cycle 2 Day 1:

Vital signs are monitored, weight is measured, perform physical examination, electrocardiogram, and ECOG score; Laboratory tests: including blood tests (hematology, blood biochemistry, coagulation function), and the required blood collection volume is about 10-20 mL; Urine routine, urine sample collection volume of approximately 10 mL; Fecal routine, stool samples are collected approximately the size of soybeans. DXC006 is administered intravenously.

Approximately 7 mL of blood samples will be collected at each blood sampling point for study drug concentration monitoring;

Cycle 2 Day 8:

Vital signs are monitored, physical examination, and ECG are performed. Laboratory tests: including blood tests (hematology, blood biochemistry, coagulation function), and the required blood collection volume is about 10-20 mL; urinalysis, urine sample collection volume is approximately 10 mL.

② Cycle 3 and subsequent cycles

Day 1:

Vital signs are monitored, weight is measured, physical examination, electrocardiogram, echocardiography, ECOG score are performed; Laboratory tests: including blood tests (hematology, blood biochemistry, coagulation function, etc.), and the required blood collection volume is about 10-20 mL; Urine routine, urine sample collection volume of approximately 10 mL; Fecal routine, stool samples are collected approximately the size of soybeans.

DXC006 is administered intravenously.

In addition, cardiac echocardiography/MUGA will be performed every 4 cycles during the study. The study doctor will also determine whether serum/urine immunofixation electrophoresis, serum free light chain, skeletal examination, extramedullary plasmacytoma test, bone marrow aspirate/biopsy, MRD assessment, CT, MRI, etc. are required based on your disease condition.

Drug concentration monitoring

Blood sampling points:

Phase 1a: within 1 h before administration, within 10 min after the end of administration, 1

 $h \pm 15$  min,  $2 h \pm 15$  min,  $6 h \pm 30$  min,  $24 h \pm 1$  h,  $72 h \pm 2$  h,  $168 h \pm 6$  h,  $240 h \pm 12$  h after the end of administration on Day 1 of Cycle 1 and Cycle 5, within 1 h before administration and within 10 min after the end of administration on Day 1 of Cycle 2; within 1 h before administration on Day 1 of Cycle 13 and every 8 subsequent cycles; once each at the end of treatment and at the safety visit. Approximately 7 mL of blood samples are collected at each time point for drug concentration monitoring.

Phase 1b: within 1 h before administration and 10 min after the end of administration in Cycles 1 and 5; within 1 h prior to administration on Day 1 of Cycle 13 and every 8 cycles thereafter; once each at the end of treatment and at the safety visit. The blood sampling time points for subjects in Phase 1b will be reasonably adjusted based on the results of previous studies. Approximately 7 mL of blood samples are collected at each time point for drug concentration monitoring.

Blood sampling for immunogenicity

Subjects will be collected once within 1 h before administration on Day 1 of Cycles 1, 3, 7, 11, 13 and every 8 cycles thereafter, at the end of treatment and at the safety visit. Survival follow-up: once every 90 days  $\pm$  7 days after the last dose. Approximately 3.5 mL of blood samples are collected at each time point for immunogenicity testing.

Metabolite identification analysis

For subjects who consent to metabolite identification are checked in the informed consent form, no separate blood sampling will be performed, and only the blood samples of spare blood will be analyzed for all drug concentration monitoring of the subjects during the clinical trial.

#### 3) End of treatment (EOT)

The End of Treatment (EOT) Visit is performed at the time the subject decides to discontinue treatment and/or withdraw from the study ( $\pm$  3 days) and the subject should go to the study site for assessments of the following items:

Vital signs are monitored, weight is measured, physical examination, electrocardiogram, and ECOG score are performed; Laboratory tests: including blood tests (hematology, blood chemistry, coagulation function, corrected serum calcium, serum protein electrophoresis, etc.), and the required blood sampling volume is approximately 10-20 mL; Urinalysis (urine routine, 24-hour urine protein electrophoresis, etc.), with a urine sample collection volume of approximately 10 mL; Fecal routine, stool samples are collected approximately the size of soybeans.

Pregnancy testing is required for women of childbearing potential and approximately 3-5 mL of blood is required.

7 mL blood sample is required for study drug concentration monitoring; 3.5 mL blood samples are collected for immunogenicity testing;

Cardiac echocardiography/MUGA is performed.

#### 4) Safety follow-up

At the Safety Follow-up Visit,  $30 \pm 7$  days after the last dose of study drug, subjects should be assessed at the study site for the following:

Vital signs are monitored, weight is measured, physical examination, electrocardiogram, and ECOG score are performed; laboratory tests: including blood tests (hematology, blood biochemistry, coagulation function), and the required blood collection volume is about 10-20 mL; Urine routine, urine sample collection volume of approximately 10 mL; Fecal routine, stool samples are collected approximately the size of soybeans.

7 mL blood sample is required for study drug concentration monitoring; 3.5 mL blood samples are collected for immunogenicity testing.

#### 5) Survival follow-up

Survival follow-up is to be performed every 90 days ( $\pm$  7 days) after the last dose to collect subject survival information (date of death and cause of death) until death, new anti-tumor therapy, or subject is lost to follow-up or discontinued from the study. Approximately 3.5 ml of blood samples are collected for immunogenicity testing.

#### 3. Other matters that require your cooperation

New information related to the study may arise during the conduct of the study project. If new information occurs, your study doctor will inform you in a timely manner and will discuss with you whether you would like to continue to participate in this study. If you decide to continue in the study, you may be asked to sign a new informed consent form. During the follow-up phase, the doctor may learn about you by telephone, outpatient follow-up, etc. If laboratory parameters or other test results are abnormal during the study, the investigator may increase the number of tests or perform further tests as clinically indicated.

#### IV. Possible Benefits of Study Participation

If you agree to participate in this study, you may not benefit, or may have disease progression, but you may also receive direct medical benefit. This product is an innovative antibody drug conjugate. Previous studies and ongoing clinical studies abroad suggest that such drugs can further improve the therapeutic efficacy of various solid tumors and hematomas such as small cell carcinoma of lung, multiple myeloma, and neuroblastoma. Your immediate benefit is that your disease may be controlled or relieved. We hope that the information obtained from

your participation in this study will be instructive in the future for patients with the same condition as you. This will provide more treatment options for cancer patients, provide clinicians with more appropriate clinical decisions, and ultimately benefit applicable patients.

# V. Possible adverse reactions, risks and discomfort, inconvenience of participating in the study

If any discomfort, or new changes in your condition, or any unexpected situation occurs during the study, whether related to the study or not, your doctor should be notified promptly, and your doctor will make a judgement about it and give appropriate medical treatment.

All drugs have adverse effects, and any study has certain risks. The study drug may contain substances that may cause you to become sick, unwell, or harmed. During your participation in the study, you may experience adverse reactions related to the study drug, as well as the risks and discomfort associated with the procedures. The study personnel will closely monitor your symptoms and adverse reactions and may give you treatments or treatments that help alleviate the adverse reactions. If the study doctor thinks you cannot tolerate these adverse reactions, study drug may be interrupted or permanently discontinued.

The effect of DXC006 on the safety of human pregnancy has not been established. General genotoxicity studies are not conducted. Therefore, DXC006 is not recommended for pregnant or lactating women. Male patients with childbearing requirements can only be enrolled if they take effective contraceptive measures during the trial and within 6 months after the end of the trial.

In addition to drug therapy, there are risks to the tests and procedures in the study, including those involved in routine medical care.

#### VI. Related costs

The investigational drug DXC006 and the investigational treatment and examination procedures mentioned in this informed consent form are all study-related. Various medical expenses related to this trial, including laboratory tests, 12-lead ECG, imaging tests, bone marrow aspirate, etc., used to evaluate safety and efficacy, will be borne by the sponsor throughout the clinical trial. The sponsor will not pay fees unrelated to this study.

You will be given certain compensation for blood sampling: including compensation for blood sampling in pharmacokinetic study: RMB 200 /blood sampling point (settlement according to the actual number of blood sampling points).

You will be given a certain amount of inpatient compensation: RMB 200 /time (settled

according to the actual number of hospitalizations). If you withdraw from the study during the study, the sponsor will compensate you for the actual number of hospitalizations.

You will be given a certain compensation fee for providing tumor tissue sections: if tumor tissue sections are provided, a subsidy of RMB 300 will be given, or RMB 1000 will be given for pathological biopsy slides.

Throughout the study period, you will be required to come to the hospital on time for follow-up as required, and the sponsor will provide transportation compensation of RMB 200/visit for these visits to the hospital (which will be settled according to the actual visit). If you withdraw from the study during the study, the sponsor will provide you with appropriate transportation compensation according to the actual number of visits.

The above fees shall be paid to you in accordance with the relevant procedures of the hospital. No compensation will be provided beyond that.

#### VII. Confidentiality of Personal Information

Your participation in the study and your personal data in the study are confidential. To protect your privacy, you will be assigned a subject number in the study. Your study doctor will keep your personal medical records and a list that links your personal medical records to your subject number. The hospital will maintain all records of you in this study and will not be accessible to any unauthorized person.

Drug regulatory authorities, ethics committees, study center staff, and representatives of the sponsor will be allowed access to these records and compare and inspect the collected study information related to you in accordance with your medical records. By signing this consent form, you allow people from these organizations to have direct access to your medical records.

The collected information may be sent to the sponsor and regulatory authorities, etc. The sponsor will use the information collected from you to publish the results of the study or to apply for registration, but will not disclose any information that identifies you personally. By signing this consent form, you agree to use your information.

You may withdraw from the study at any time, but if permitted by law, the sponsor will continue to use the information collected prior to your withdrawal.

### VIII. How to get more information?

You may ask any questions about this study at any time during the study. Your study doctor will leave you his/her telephone number so that you can answer your questions.

Your study doctor will notify you in a timely manner if there are any important updates to

information during the study that may affect your willingness to continue in the study. We will modify the contents of the informed consent form and will be re-signed and confirmed by you or your legal representative.

#### IX. May voluntarily choose to participate in the study and withdraw from the study

Your participation in this study is entirely voluntary. You may choose not to participate in this study without being affected, discriminated against, retaliated, or compromised; even if you agree to participate in this study, you may withdraw from the study at any time for any reason, you will not be discriminated against or retaliated for withdrawing from the study, and your normal medical treatment will not be affected in any way. If you withdraw from the study for any reason, you are expected to inform your study doctor in a timely manner, who can provide advice and guidance on your health.

The doctor or investigator may stop you from continuing in this study at any time during the study for the best interests of you.

#### X. What should you do now?

It is up to you (and your guardian) to decide whether to take part in this study.

Ask your doctor as many questions as possible before you make your decision to participate in the study.

Thank you for reading the above materials. If you decide to take part in this study, tell your doctor that he/she will take care of you of all study-related matters. This informed consent form is provided in duplicate, one for the subject and one for the investigator, and is valid for signature by both parties. You will be given an original signed and dated informed consent form.

### Informed consent. Consent Signature Page

| A Phase 1, Open-label, Multi-center, First-in-Human, Dose | |
|---|---|
| Escalation and Expanded-enrollment Clinical Study to Evaluate | |
| the Safety, tolerability, Pharmacokinetic Characteristics and | |
| Preliminary Efficacy of DXC006 for Injection in Patients with | |
| Multiple Solid Tumors and Hematomas | |
| The Cancer Center of Sun Yat-sen University N/A | |
| | DAC000-001 |

#### **Statement of Consent**

I have read the above description of this study and have had the opportunity to discuss and ask questions with my doctor about this study. All my questions are answered to my satisfaction.

I am aware of the risks and benefits that may arise from taking part in this study. I am aware that participation in the study is voluntary and I confirm that there is sufficient time to consider this and understand that:

- I can ask my doctor for more information at any time.
- I can withdraw from this study at any time without discrimination or retaliation, and medical treatment and rights will not be affected.

I am also aware that if I withdraw from the study halfway, especially if I am withdrawn from the study due to drug reasons, it will be very beneficial for the entire study if I inform the doctor of my condition changes and complete the corresponding physical and physical and chemical examinations.

If I need to take any other medication due to a change in my condition, I will consult my doctor in advance, or tell the doctor truthfully afterwards.

I agree that the Ethics Committee of the drug regulatory authority or the sponsor's representative shall have access to my study data.

I will receive an original signed and dated informed consent form.

Finally, I decided to agree to participate in this study and to ensure that my doctor's instructions are followed as much as possible, and that I did not participate in other clinical studies during this study.

| Patient Signature: | Year _ | _Month _ | _Day |
|--------------------|--------|----------|------|
| Tel: | | | |

I confirm that the details of this trial, including their rights and possible benefits and risks, have been explained to the patient and a copy of the signed informed consent form has been given to the patient.

| DXC006 | Hangzhou DAC Biotechnology Co., Ltd. |
|-----------------------------|--------------------------------------|
| Doctor Signature: | YearMonthDay |
| Doctor's Work Phone Number: | _ |